CLINICAL TRIAL: NCT05650749
Title: Phase 1 Trial of GPC2-Directed Chimeric Antigen Receptor Autologous T Cells (GPC2 CAR T) for Relapsed or Refractory Neuroblastoma and Metastatic Retinoblastoma
Brief Title: GPC2 CAR T Cells for Relapsed or Refractory Neuroblastoma and Metastatic Retinoblastoma
Acronym: GPC2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Gilead Sciences (Industry); University of Pennsylvania (Other); National Cancer Institute (NCI) (NIH); Kite, A Gilead Company (Industry)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Chief, Cell Therapy and Transplant Section Director, Susan S. and Stephen P. Kelly Center for Cancer Immunotherapy Medical Director, Cell and Gene Therapy Lab, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-019659; 1R37CA282041-01A1 (NIH); 22CT012 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Refractory Neuroblastoma; Relapsed Neuroblastoma; High-risk Neuroblastoma; Retinoblastoma; Metastatic Retinoblastoma
MeSH Terms: conditions — Neuroblastoma; Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Arm (Experimental): The dose escalation arm will determine the maximum tolerated dose of GPC2 CAR T cells using a standard 3+3 trial design.
  Interventions: Biological: GPC2 CAR T cells
- Dose Expansion Arm (Experimental): If at least one dose from the dose expansion arm is determined to be safe, additional patients will be enrolled to the dose expansion arm to preliminarily evaluate the rate of response to GPC2 CAR T cells and further characterize the safety profile of GPC2 CAR T cells.
  Interventions: Biological: GPC2 CAR T cells

INTERVENTIONS:
Biological: GPC2 CAR T cells — The GPC2 CAR T investigational product is comprised of autologous human T cells that have been genetically modified to express a GPC2-targeting chimeric antigen receptor (CAR) transgene.

SUMMARY:
This is a first in human dose escalation trial to determine the safety of administering GPC2 CAR T cells in patients with advanced neuroblastoma or retinoblastoma.

DETAILED DESCRIPTION:
Despite the use of intensive multimodal chemoradiotherapy, surgery, autologous stem cell transplant and GD2-targeted immunotherapy for the treatment of patients with high-risk neuroblastoma, approximately 60% of children still die from this disease and survivors suffer lifelong treatment related comorbidities. Similarly, children with retinoblastoma with extra-ocular metastasis experience a poor prognosis despite the availability of intensive systemic chemotherapy or external beam radiation therapy. Among children with metastatic retinoblastoma treated with intensive multimodality treatment, 3-year Event Free Survival ranges from 14 to 77% depending on central nervous system (CNS) involvement. For neuroblastoma and retinoblastoma patients who suffer a relapse after receiving therapy with standard of care multimodality treatment, there are no known curative options. Glypican 2 (GPC2) is highly expressed on the plasma membrane of most high-risk neuroblastomas and retinoblastomas, is further enriched in the tumor stem cell compartment, but is not expressed at significant levels on normal tissues, making it an ideal target for immune directed therapies. To therapeutically leverage GPC2's differential expression, we have developed a GPC2-directed CAR T cell therapy that potently inhibits the growth of neuroblastoma and retinoblastoma patient-derived xenografts. This investigation will be a single institution, open label first in human, dose escalation and expansion study designed to assess the safety, tolerability, and manufacturing feasibility of GPC2 CAR T cells.

ELIGIBILITY:
Neuroblastoma Inclusion Criteria:

1. Patients must be ≥ 1 year of age
2. Patients must have high-risk neuroblastoma according to COG risk classification at the time of study enrollment. Patients who were initially considered low- or intermediate-risk, but then reclassified as high-risk are also eligible.
3. Patients must have a previously histologically confirmed diagnosis of neuroblastoma:

   1. That is recurrent/relapsed or refractory/persistent according to INRC AND
   2. For which standard curative measures do not exist or are no longer effective.
   3. patients at first relapse are eligible as no known curative therapies exist for relapsed high-risk neuroblastoma.
4. Patients must have evaluable or measurable disease at enrollment.
5. In addition, patient must have experienced at least one of the following:

   a. New disease site documented on at least one of the following: i. 123I-meta-iodobenzylguanidine (MIBG) or 18F-mFBG (meta-fluorobenzylguanidine) scan; OR ii. CT/MRI; OR iii. FDG or Ga-68 Dotatate PET (in patients known to have MIBG non-avid tumor) and MRI findings consistent with tumor (i.e., bone lesions), OR iv. Biopsy confirmed neuroblastoma for any new or progressing lesion. b. Greater than 20% increase in a least one dimension of soft tissue mass documented by CT/MRI and a minimum absolute increase of 5 mm in longest dimension in existing lesion(s). Previously irradiated lesions may be included.

   c. Bone marrow biopsy shows progressive disease according to the revised INRC d. Stable persistent disease, such that response at the completion of upfront therapy or salvage therapy is less than partial response AND has a biopsy of at least one site showing viable neuroblastoma.

   e. Responding persistent disease, defined as at least a partial response to frontline therapy (i.e., at least a partial response to frontline therapy but still has residual disease by MIBG scan, CT/MRI, or bone marrow aspirations/biopsies). Patients in this category are required to have histologic confirmation of viable neuroblastoma from at least one residual site (tumor seen on routine bone marrow morphology is sufficient).
6. Patients must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of ≥ 60
7. Patients must have adequate renal function defined as age-adjusted serum creatinine ≤1.5 ULN for age.
8. Total bilirubin ≤ 1.5 x ULN (exception: total bilirubin ≤ 3 ULN for patients with Gilbert's Disease)
9. Aspartate aminotransferase (AST) ≤ 2.5 ULN (exception: AST ≤ 5 x ULN for patients with liver metastases).
10. Alanine aminotransferase (ALT) ≤ 2.5 ULN (exception: ALT ≤ 5 x ULN for patients with liver metastases).
11. Patients must have a baseline pulse oximetry of at least 92% on room air. In addition, a DLCO ≥ 60% (corrected for anemia) is required if PFTs are clinically appropriate as determined by the treating investigator.
12. Left ventricular shortening fraction (LVSF) ≥28% or ejection fraction (LVEF) ≥ 50% confirmed by Echo, or adequate ventricular function documented by a scan or a cardiologist.

Neuroblastoma Exclusion Criteria:

1. Patients with active hepatitis B or active hepatitis C.
2. Patients with HIV infection.
3. Patients with uncontrolled active infection.
4. Patients with primary or acquired immunodeficiency disorder.
5. Patients with a known hypersensitivity to DMSO.
6. Concurrent use of systemic steroids or immunosuppression at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy or immunosuppression during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
7. Patients with actively progressing CNS metastases, including parenchymal or leptomeningeal involvement. (Note: CNS imaging at screening is only required if the there is a clinical indication of suspected CNS metastasis)
8. Active medical disorder that, in the opinion of the investigator, would substantially increase the risk of uncontrollable CRS and/or neurotoxicity.
9. Patients with congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis.
10. Patients who have received any live vaccines within 30 days prior to enrollment.
11. Patients who are pregnant or nursing (lactating).
12. Patients who have a life expectancy < 6 months at time of consent.

Retinoblastoma Inclusion Criteria:

1. Patient age ≥ 6 months.
2. Patients must have metastatic retinoblastoma according to International

   Retinoblastoma Staging System (IRSS) risk classification (4) at the time of study enrollment:

   a. Retinoblastoma Cohort 1 (Extra-CNS metastasis) i. Stage IVa disease ii. Extra-CNS disease must be confirmed as retinoblastoma by histology (either at diagnosis or recurrence) iii. Measurable disease: Defined as > 1cm2 or biopsy-proven bone marrow disease iv. Prior treatment: Recurrent or refractory disease following treatment with COG ARET0321-like or equivalent regimen as part of upfront or recurrent therapy b. Retinoblastoma Cohort 2 (CNS disease) i. Stage IVb disease ii. Histologic confirmation is not required iii. CNS disease defined as measurable disease >1cm2, non-measurable, or CSF positivity alone c. Prior treatment: i. Stage IVb.1 and IVb.2: Recurrent after treatment with COG ARET0321-like or equivalent regimen as part of upfront or recurrent therapy i. Stage IVb.3: Prior treatment is not required (i.e., eligible at initial diagnosis or recurrence)
3. Patients must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of ≥ 60
4. Patients must have adequate renal function defined as age-adjusted serum creatinine ≤1.5 ULN .
5. Total bilirubin ≤ 1.5 x ULN (exception: total bilirubin ≤ 3 ULN for patients with Gilbert's Disease)
6. Aspartate aminotransferase (AST) ≤ 2.5 ULN (exception: AST ≤ 5 x ULN for patients with liver metastases).
7. Alanine aminotransferase (ALT) ≤ 2.5 ULN (exception: ALT ≤ 5 x ULN for patients with liver metastases).
8. Patients must have a baseline pulse oximetry of at least 92% on room air. In addition, a DLCO ≥ 60% (corrected for anemia) is required if PFTs are clinically appropriate as determined by the treating investigator.
9. Left ventricular shortening fraction (LVSF) ≥28% or ejection fraction (LVEF) ≥ 50% confirmed by Echo, or adequate ventricular function documented by a scan or a cardiologist.

Retinoblastoma Exclusion Criteria:

1. Patients with active hepatitis B or active hepatitis C.
2. Patients with HIV infection.
3. Patients with uncontrolled active infection.
4. Patients with primary or acquired immunodeficiency disorder.
5. Patients with a known hypersensitivity to DMSO.
6. Concurrent use of systemic steroids or immunosuppression at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy or immunosuppression during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
7. Active medical disorder that, in the opinion of the investigator, would substantially increase the risk to the subject.
8. Patients with congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis.
9. Patients who have received any live vaccines within 30 days prior to enrollment.
10. Patients who are pregnant or nursing (lactating).
11. Patients who have a life expectancy < 6 months at time of consent.
12. Retinoblastoma Cohort 1 (Extra-CNS disease):

    1. Concurrent CNS disease (they may be eligible for Retinoblastoma Cohort 2)
    2. Stage III disease (orbital or lymph node regional extension without other hematogenous metastases).
13. Retinoblastoma Cohort 2 (CNS disease):

    1. "Bulky" disease (>5 cm in diameter) within or compressing the brainstem or thalamus. Note: Tumors touching the brainstem/thalamus without evidence of compression and/or tumors in other CNS locations do not have a maximal size criterion.
    2. If evidence of clinically significant increased intracranial pressure at time of relapse, patient must demonstrate improvement by time of enrollment.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose of GPC2 CAR T cells | 5 years
  The Maximum Tolerated Dose of GPC2 CAR T cells will be determined by measuring the incidence of dose limiting toxicities following administration of the product.
Frequency of Adverse Events Following GPC2 CAR T cell administration | 5 years
  Assess the frequency and severity of treatment related adverse events following administration of GPC2 CAR T cells.

SECONDARY OUTCOMES:
Manufacturing Feasibility of GPC2 CAR T cells | 5 years
  Manufacturing Feasibility will be evaluated as the Percentage of patients with GPC2 CAR T cell products that meet release criteria
Persistence of GPC2 CAR T cells | 5 years
  Persistence of GPC2 CAR T cells will be measured by Polymerase Chain Reaction (or flow cytometry) analysis of whole blood to detect and quantify survival of GPC2 CAR T cells over time.
Preliminarily define the clinical activity of GPC2 CAR T in patients with relapsed or refractory neuroblastoma or metastatic retinoblastoma | 5 years
  Overall Response Rate will be determined based on international Neuroblastoma Response Criteria or the COG Retinoblastoma ARET0321/ Response and Response Assessment in Pediatric Neuro-Oncology.
Severity of Adverse Events Following GPC2 CAR T cell administration. | 5 years
  The safety of GPC2 CAR T cell therapy reinfusions will be measured by the monitoring the frequency and severity of adverse events after multipleGPC2 CAR T cells infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wray, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giudice AM, Matlaga S, Roth SL, Gladney W, Groff D, Hofmann TJ, McDaid KS, Pascual-Pasto G, McIntyre B, Zecchino V, Martinez D, Spear TT, Wolpaw AJ, Assenmacher CA, Radaelli E, Pogoriler J, Pawel B, Barrett D, Grupp SA, Maris JM, Bosse KR. D3-GPC2-Directed CAR T Cells Are Safe and Efficacious in Preclinical Models of Neuroblastoma and Small Cell Lung Cancer. Clin Cancer Res. 2025 Dec 15;31(24):5276-5293. doi: 10.1158/1078-0432.CCR-25-0089. PMID 41026583